CLINICAL TRIAL: NCT01636830
Title: The Incidence of Gingival Fissures _ a Crossover Single-blinded Randomized
Brief Title: The Incidence of Gingival Fissures _ a Crossover Single-blinded Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Bruna Frizon Greggianin, Rui Vicente Oppermann, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BR 001
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Gingival Recession; Wounds and Injuries
Keywords: Toothbrushing; gingival recession
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toothbrush type - medium (Active Comparator): This is a crossover study, where the person used either a soft brush (control) and the medium brush (test).
  Interventions: Device: Toothbrush type
- Toothbrush type - soft (Active Comparator): This is a crossover study, where the person used either a soft brush (control)and the medium brush(test).
  Interventions: Device: Toothbrush type

INTERVENTIONS:
Device: Toothbrush type — Evaluate the use of toothbrushes with bristles soft and medium

SUMMARY:
The objective of this study is to evaluate the incidence of gingival fissures according to the type of brush used, soft and medium.

DETAILED DESCRIPTION:
Gingival recession constitute a functional and aesthetic problem that affects much of the population. One of the possible causes refers to a traumatic brushing. Individuals who have an excessive tooth brushing can cause injuries to your gums, such as abrasions and fissures. These lesions have been considered subrogated outcomes of gingival recession noninfectious. The literature only reports and case series showing the gingival fissures, which were once associated with traumatic occlusion.

This is the first clinical trial to evaluate the gingival fissures according to the type of brush used.

ELIGIBILITY:
Inclusion Criteria:

* good/ excellent health;
* idade de 14 a 20 anos;
* at least 20 teeth without a history of destructive periodontal disease, absence of gingival bleeding;
* absence of loss of attachment/recession ≥2mm in molars and pre-molars in the buccal areas.

Exclusion Criteria:

* were unable to provide consent or comply with the sudy protocol;
* smokers;
* pregnant women;
* persons under orthodontic treatment or with dental or implant prosthesis, presence of cervical abrasions, restorations or caries;
* need of antibiotic prophylaxis associated with dental procedures.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Gingival Fissures associated with toothbrushing | 3 months
  This study took standardized photographs every 2 or 3 days during two periods of 28 days for evaluation of gingival fissures. These were measured by application of a disclosing solution of plaque on teeth and gums of the participants. The application developer board is safe, without contra-indications in the literature and facilitates visualization of gingival lesions and plaque.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Greggianin BF, Oliveira SC, Haas AN, Oppermann RV. The incidence of gingival fissures associated with toothbrushing: crossover 28-day randomized trial. J Clin Periodontol. 2013 Apr;40(4):319-26. doi: 10.1111/jcpe.12072. Epub 2013 Feb 21. PMID 23425194
- See also: Website of the Federal University of Rio Grande do Sul — http://www.ufrgs.br/odonto